CLINICAL TRIAL: NCT02993965
Title: State Immunization Information Systems to Improve HPV Vaccination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, Los Angeles (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 15-1560; 1R01CA187707-01A1 (NIH)
Record Dates: First submitted 2016-11-29; First posted 2016-12-15 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Vaccine; Human Papiloma Virus Vaccine; HPV Vaccine; Immunization; Health Registry; Adolescent Health; Reproductive Health; Preventive Health Services

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control 11-17 (No Intervention): No additional intervention done aside from usual care for 11-17 year olds
- 1 R/R per Dose 11-17 (Experimental): Sending up to one recall notice per dose of HPV vaccine needed for 11-17 year olds
  Interventions: Other: Vaccine Reminder/Recall
- 2 R/R per Dose 11-17 (Experimental): Sending up to two recall notices per dose of HPV vaccine needed for 11-17 year olds
  Interventions: Other: Vaccine Reminder/Recall
- 3 R/R per Dose 11-17 (Experimental): Sending up to three recall notices per dose of HPV vaccine needed for 11-17 year olds
  Interventions: Other: Vaccine Reminder/Recall
- Control 11-14 (No Intervention): No additional intervention done aside from usual care for 11-14 year olds
- Phone R/R 11-14 (Experimental): Sending up to two recall notices per dose of HPV vaccine needed via autodialer for 11-14 year olds
  Interventions: Other: Vaccine Reminder/Recall
- Mail R/R 11-14 (Experimental): Sending up to two recall notices per dose of HPV vaccine needed via mailed postcards for 11-14 year olds
  Interventions: Other: Vaccine Reminder/Recall

INTERVENTIONS:
Other: Vaccine Reminder/Recall — The investigators will be sending recall notices via phone call or postcard to 11-17 year olds or 11-14 year olds who are eligible but lacking HPV vaccine doses recorded in the Colorado Immunization Information System (CIIS). The investigators will be testing the effectiveness and cost effectiveness of up to 3 notices per dose with usual care (no intervention) for bringing children 11-17 years old up to date on HPV vaccination. They will also be testing the effectiveness and cost effectiveness of using mail vs. phone call reminder notices (as compared to no intervention) for bringing 11-14 year olds up to date on HPV vaccination.
  Arms: 1 R/R per Dose 11-17; 2 R/R per Dose 11-17; 3 R/R per Dose 11-17; Mail R/R 11-14; Phone R/R 11-14

SUMMARY:
The overarching goal of this study is to evaluate the effectiveness, cost-effectiveness and sustainability of utilizing statewide Immunization Information Systems (IIS) to conduct centralized reminder/recall (R/R) to improve Human Papiloma Virus (HPV) vaccination rates among adolescents ages 11-17 (with a more focused look at the new two dose series for 11-14 year olds).

DETAILED DESCRIPTION:
The overarching goal of this study is to evaluate the effectiveness, cost-effectiveness and sustainability of utilizing statewide Immunization Information Systems (IIS) to conduct centralized reminder/recall (R/R) to improve HPV vaccination rates among adolescents ages 11-17, and additionally look at the 11-14 year old subset for whom a new 2 dose series has recently been recommended. The investigators will extend previous research on effectiveness of centralized R/R to a new population--adolescents due for HPV vaccine-- and test the use of centralized R/R as a cancer-prevention strategy. Investigators will assess the effect of centralized R/R in two states--one with and one without mandated reporting of vaccinations to IISs, and disseminate IIS R/R to other states. Investigators will implement, evaluate (using the RE-AIM framework 31-36), and disseminate a collaborative, IIS-based centralized HPV vaccine R/R model in which partnerships of public health systems and primary care practices in two states (NY, CO) collaborate to remind parents about HPV vaccination.

Specific Aims and hypotheses:

Aim #1: Adapt IIS messages and delivery systems (e.g., algorithms) previously developed for centralized R/R for other vaccines to fit HPV vaccine IIS R/R.

Aim #2: Assess the impact and cost-effectiveness of centralized IIS-based (IIS-C) autodialer (phone) R/R in increasing vaccine rates [initial dose (HPV#1) and a complete series (HPV#2 or #3)] among teens.

Conduct a pragmatic trial, to assess the impact and cost effectiveness of centralized IIS-based (IIS-C) autodialer (phone) R/R in increasing initiation and completion rates for the HPV vaccine series in adolescents ages 11-17 years. The investigators will use a within-practice design, randomizing patients within randomly selected primary care practices to IIS-C R/R (1, 2, or 3 reminders per dose) compared to usual care (0 reminders from this study). The investigators will apply the RE-AIM framework to evaluate the reach, effectiveness/cost effectiveness, adoption, and implementation of IIS-C R/R.

Hypothesis 2a: IIS-C R/R will result in higher HPV vaccination rates than usual care.

Hypothesis 2b: IIS-C R/R will result in higher HPV vaccination rates than usual care in key subgroups (males and females, younger and older teens, urban//rural teens).

Hypothesis 2c: IIS-C R/R will be more cost-effective (cost/vaccine received) than usual care.

Aim #3: Assess the impact and cost-effectiveness of centralized IIS-based (IIS-C) R/R using autodialer (phone) or mail in increasing vaccine rates [initial dose (HPV#1) and a complete series (HPV#2)] and decreasing time to completion among teens 11-14.

Conduct a pragmatic trial, to assess the impact and cost effectiveness of centralized IIS-based (IIS-C) R/R using either autodialer (phone) or postcard (mail) in increasing initiation and completion rates for the newly implemented HPV vaccine 2 dose series in adolescents ages 11-14 years. We will use a within-practice design, randomizing patients within randomly selected primary care practices to IIS-C R/R using either an autodailer or postcards (up to 2 reminders per dose needed) compared to usual care (0 reminders from this study). We will apply the RE-AIM framework to evaluate the reach, effectiveness/cost effectiveness, adoption, and implementation of IIS-C R/R.

Hypothesis 3a: IIS-C R/R (either modality) will result in higher HPV vaccination rates than usual care.

Hypothesis 3b: IIS-C R/R (either modality) will result in higher HPV vaccination rates than usual care in key subgroups (males and females, younger and older teens, urban//rural teens).

Hypothesis 3c: IIS-C R/R will be more cost-effective (cost/vaccine received) than usual care. IIS-C R/R using autodialer will be more cost effective than IIS-C R/R using postcards.

Aim #4: Disseminate IIS-C R/R across NY and CO and pilot in four IISs: (a) Develop an IIS-C HPV R/R toolkit, (b) Use a technical advisory group, (c) Initiate IIS-C R/R in four other IISs [Yr. 4].

By the end of the study investigators will have a feasible, sustainable, cost-effective model for HPV vaccine reminders that can be used nationally to prevent cervical cancer and other HPV-related cancers.

ELIGIBILITY:
Inclusion Criteria:

* 11 through 17 years of age (trial 1)
* 11 through 14 years of age (trial 2)
* defaulted to our selected clinics within CIIS
* is either due for an HPV dose at baseline according to Advisory Committee on Immunization Practices (ACIP) guidelines, or
* has initiated but not yet completed the HPV series at baseline

Exclusion Criteria:

* Has completed the HPV vaccine series according to Advisory Committee on Immunization Practices (ACIP) guidelines
* Any child whose parents have requested removal from the immunization registry

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77716 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Initiation of the HPV vaccine series (receipt and documentation of initial dose of vaccine series within immunization registry) | 5 months
  Did the adolescent initiate the HPV vaccine series? The investigators are allowing up to 5 months after the initial recall notice for the adolescent to make an appointment and receive their dose. After that time frame, the investigators will not attribute vaccination to the recall. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry.
Completion of the HPV vaccine series (receipt and documentation of final dose of vaccine series within immunization registry) | 5 months
  Did those eligible to complete the HPV vaccine series within the time frame of the study do so? The investigators are allowing up to 5 months after the initial recall notice for the adolescent to make an appointment and receive their dose. After that time frame, the investigators will not attribute vaccination to the recall. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry.

SECONDARY OUTCOMES:
Differences between arms - initiation | 5 months
  Is 1, 2, or 3 reminders per arm most effective and cost effective for initiation. Only those who need an initial dose at baseline will be eligible for this outcome. Adolescents in each arm will be allowed up to 5 months after the first recall notice to get a vaccine. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry. This will be tested in the 11-17 year old group.
Differences between arms - completion | 20 months
  Is 1, 2, or 3 reminders per arm most effective and cost effective for completion. Because the second or third dose of the series is dependent on when the adolescent receives their initial dose, the investigators will be following eligible adolescents for 20 months to allow time for those who did not respond to the recall for the initial dose right away to be able to complete the series within the time frame. However, receipt of the completion dose will only be attributed to the recall if it was received within 5 months of the 1st recall for the completion dose. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry. This will be tested in the 11-17 year old group. For 11-14 year olds, completion is 2 doses. For 15-17 year olds, completion is 3 doses.
Differences between modalities - initiation | 5 months
  Are mail or phone reminders most effective and cost effective for initiation. Only those who need an initial dose at baseline will be eligible for this outcome. Adolescents in each arm will be allowed up to 5 months after the first recall notice to get a vaccine. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry. This will be tested with the 11-14 year old group only.
Differences between modalities - completion | 5 months
  Are mail or phone reminders most effective and cost effective for completion. This will be tested only in the 11-14 year old group, so completion will equal 2nd dose. Because the second dose of the series is dependent on when the adolescent receives their initial dose, the investigators will be following eligible adolescents for 17 months to allow time for those who did not respond to the recall for the initial dose right away to be able to complete the series within the time frame. However, receipt of the completion dose will only be attributed to the recall if it was received within 5 months of the 1st recall for the completion dose. Receipt will be documented by providers within the state immunization registry via EMR direct transfer or manual entry.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual data with other researchers

REFERENCES:
- [Derived] Gurfinkel D, Kempe A, Albertin C, Breck A, Zhou X, Vangala S, Beaty B, Rice J, Tseng CH, Campbell JD, Valderrama R, Rand C, Humiston SG, Roth H, Arora S, Szilagyi P. Centralized Reminder/Recall for Human Papillomavirus Vaccination: Findings From Two States-A Randomized Clinical Trial. J Adolesc Health. 2021 Oct;69(4):579-587. doi: 10.1016/j.jadohealth.2021.02.023. Epub 2021 Apr 10. PMID 33846054